CLINICAL TRIAL: NCT01294215
Title: A Multicenter, Open Label, Long Term Study of Oral BAYA1040_CR 80 mg (40 mg Bid) in Combination With Other Antihypertensives for 52 Weeks in Patients With Essential Hypertension
Brief Title: High Dose BAYA1040_Nifedipine: a Long Term Combination Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14024
Record Dates: First submitted 2011-02-10; First posted 2011-02-11 (Estimated); Last update posted 2014-06-23 (Estimated); Status verified 2014-06

CONDITIONS: Hypertension
Keywords: BAYA1040; Nifedipine; Essential hypertension; Japanese Patients; Phase III; combination study; 14024
MeSH Terms: conditions — Hypertension; Essential Hypertension | interventions — Nifedipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Nifedipine (Adalat, BAYA1040)

INTERVENTIONS:
Drug: Nifedipine (Adalat, BAYA1040) — Nifedipine (Adalat, BAYA1040) 40mg twice a day (BID)

SUMMARY:
This is a clinical study evaluating the safety and efficacy of long term administration of oral BAYA1040_Nifedipine 80 mg/day (40 mg twice daily) with other antihypertensives in patients with essential hypertension who are not at target blood pressure by the combination of BAYA1040_Nifedipine 40 mg once daily and other antihypertensives.

ELIGIBILITY:
Inclusion Criteria:

* 20 years or older
* Japanese male or female
* Outpatient with essential hypertension
* Patients who are treated with Adalat CR 40 mg od and at least one antihypertensive drug (other than Ca antagonists) for 4 weeks or more before entry in this study

Exclusion Criteria:

* Patients whose sitting diastolic blood pressure (DBP) is 110 mm Hg or more
* Patients with secondary hypertension or hypertensive emergency

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2011-02; Primary Completion 2011-11 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Efficacy changes measured by sitting diastolic blood pressure (DBP) | Up to 52 weeks

SECONDARY OUTCOMES:
Efficacy changes measured by sitting systolic blood pressure (SBP) | Up to 52 weeks
Proportion of subjects achieving a target BP based on the Japanese Society of Hypertension (JSH) 2009 guidelines | Up to 52 weeks
Proportion of subjects achieving a target DBP and SBP based on JSH 2009 guidelines or a >10 mmHg reduction of DBP | Up to 52 weeks
Safety variables | Up to 30 days after the last dose of study drug
  Adverse events, vital signs, electrocardiography (ECG), and laboratory tests were evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (4):
- Japan (4):
  - Ebina, Kanagawa
  - Sagamihara, Kanagawa
  - Kawaguchi, Saitama
  - Shinjuku, Tokyo